CLINICAL TRIAL: NCT07365293
Title: Testing Implementation Strategies to Scale-up a Multicomponent Continuum of Service Intervention for Families Involved in Systems With Parental Opioid and Methamphetamine Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Saldana, Research Scientist, Chestnut Health Systems
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-60; RM1DA064527 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Substance Related Disorders
Keywords: opioid; child welfare; prevention; evidence-based; implementation; stimulants
MeSH Terms: conditions — Substance-Related Disorders | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: Ongoing delivery of JCFF in active counties supports commencement of recruitment upon IRB approval in Year 1. Eligible parents in new counties will be recruited as a no-treatment Usual Services control in Year 1. In Year 2, both active and new clinics will be assigned to two groups, balanced by county social risk factors and child welfare outcomes, and "stepped" from their Year 1 condition to receive JCFF with the addition of the JCFF App (JCFF+ App), and then again, when FB is provided to Coaches (JCFF+App+FB). Parents will be assigned to one of four conditions: JCFF, JCFF + a digital App alone, JCFF + the App and intervention Coach feedback (FB) or usual services. Thus, intervention condition varies over time for counties, teams, and Coaches, but it is a single status for each parent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention (No Intervention): No services will be offered to participants. Participants are able to engage in any non-Just Care services that they choose, which could include substance use treatment, mental health treatment, child welfare or self-sufficiency case plans that include parenting classes, social services to access basic needs like food stamps, and support to obtain employment. Just Care for Families is not available in the counties during usual services recruitment.
- Just Care for Families (JCFF) only (Experimental): Just Care for Families is a behavioral intervention to address the needs of families involved in or at-risk for involvement with the child welfare system.
  Interventions: Behavioral: Just Care for Families (JCFF)
- Just Care for Families (JCFF) plus App (Experimental): Participants will receive the Just Care for Families (JCFF) behavioral intervention in addition to using a JCFF digital support application (App).
  Interventions: Behavioral: Just Care for Families (JCFF); Behavioral: Just Care for Families (JCFF) App
- Just Care for Families (JCFF) plus App plus Feedback (Experimental): Participants will receive the Just Care for Families (JCFF) behavioral intervention, use of the App, and the intervention coaches will receive feedback on parent's use of the App.
  Interventions: Behavioral: Just Care for Families (JCFF); Behavioral: Just Care for Families (JCFF) App; Behavioral: Just Care for Families (JCFF) App Feedback

INTERVENTIONS:
Behavioral: Just Care for Families (JCFF) — Just Care for Families is a behavioral intervention to address the needs of families involved in or at-risk for involvement with the child welfare system. Just Care involves treatment components, supported by ongoing purposeful engagement: (1) Substance use treatment including contingency management and positive reinforcement, day planning, healthy environments and peer choices, and refusal skills; (2) Mental health treatment including cognitive behavioral therapy, developing healthy coping skills, emotion regulation skills, exposure therapy, and referral for medication management; (3) Parent management training including parenting skills, nurturing and attachment, reinforcement, emotion regulation, supervision, structure, non-harsh discipline, and nutrition; (4) Community building including indigenous and external social supports; (5) Systems navigation; and (6) provision of assistance with basic needs including assistance with housing and employment.
  Arms: Just Care for Families (JCFF) only; Just Care for Families (JCFF) plus App; Just Care for Families (JCFF) plus App plus Feedback
Behavioral: Just Care for Families (JCFF) App — Participants will use a Just Care for Families digital support application (App). App features will include interactive tools modeled after those used for in-person interventions and practice exercises. Parent data will be stored within the App, including entered self-report and usage data.
  Arms: Just Care for Families (JCFF) plus App; Just Care for Families (JCFF) plus App plus Feedback
Behavioral: Just Care for Families (JCFF) App Feedback — Coaches will receive feedback on parent's use of the App. Parent-reported current needs, clinical status (e.g., substance use and mental health symptoms), progress, and goals will be programmed into dashboards accessible to assigned Coaches (i.e., Feedback).
  Arms: Just Care for Families (JCFF) plus App plus Feedback

SUMMARY:
This study will explore how to expand the Just Care for Families (JCFF) program beyond its current sites in Oregon, while addressing two main challenges: the developer team cannot provide ongoing support to every new program, and rural counties face limits on caseloads and reimbursement because of long travel distances. To overcome these barriers, the trial will test two strategies-using a JCFF mobile app to improve outcomes and efficiency, and relying on trained Experts (instead of the developer team) to guide new counties. With five active counties and four new ones, researchers will study whether parents receiving JCFF with digital support show reduced opioid and stimulant use, better child welfare outcomes like reunification, and more efficient treatment. This study will also compare how well new counties implement JCFF compared to existing ones, and use modeling to see if digital tools help programs sustain themselves by balancing caseloads and reimbursement.

DETAILED DESCRIPTION:
This Hybrid Type II effectiveness-implementation trial uses an adaptation of a stepped-wedge design to test clinical outcomes spanning interception points within the Child Welfare system and implementation outcomes when Just Care for Families (JCFF) is delivered with the addition of a mobile App with provider feedback about parent App usage. Nine rural Oregon counties, five active counties previously implemented with developer support, and four new counties that will implement with new JCFF Expert support have been recruited to test the clinical effectiveness of JCFF when delivered with and without the App. A total of 254 parents with opioid and/or stimulant use and intersection with the Child Welfare system will be recruited to participate. Parents will receive usual services, JCFF, JCFF with the App, or JCFF with the App and feedback. Longitudinal in-person assessments at baseline, 4-months, 9-months, 14-months, and 18-months, and weekly text assessments of social determinants of health needs and Child Welfare intersection will test the reduction in parent opioid and stimulant use over time with increased treatment engagement, retention, completion and decreased length of Child Welfare case, reentry into treatment, and recidivism (arrest, Child Welfare re-referral). The effectiveness of the JCFF implementation approach will be tested when implemented with the support of new JCFF Experts versus developer Experts, with the aim of equal effectiveness. Clinical and implementation outcomes will be modeled to examine the impact that adding the App could have on program sustainment for rural programs, expanding the potential for JCFF to scale up in Oregon and elsewhere, positioning for public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Misuse of opioids and/or stimulants in the last year, including misuse of prescriptions
* parent of a child aged 0-18 with the child living in the home or a reunification plan in place
* residing in one of the nine participating counties
* insured by Medicaid
* access to a computer, smartphone, or wireless/cellular connection if a device were to be provided
* Willing to enroll with the first available Just Care coach

Exclusion Criteria:

-- Alcohol use disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Opioid and/or Stimulant Use from Baseline to 18 months | Baseline, 4 months, 9 months, 14 months, and 18 months
  Any opioid or stimulant use in the past 30 days as measured by the Addiction Severity Index.
Treatment Engagement | Up to 18 months
  Number of sessions attended as reported by coaches in the Just Portal software used as part of the JCFF delivery and fidelity monitoring.
Treatment Retention | Up to 18 months
  Retained in treatment through completion (i.e. mutual decision between client and coach for how to end treatment). Measured only for the first treatment episode.
Child Welfare Re-Report | Up to 18 months
  Any new referrals for parent or child as reported in Oregon Department of Human Services Administrative Data.

SECONDARY OUTCOMES:
Child Reunification | Up to 18 months
  Any record of child being reunified with parent as reported in Oregon Department of Human Services Administrative Data.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD except for administrative data will be shared. For administrative data, a data use agreement signed by the research team and members of the third party will define the scope of appropriate access and use of the data. While overall or composite scores may be available to share publicly, ethical and legal considerations limit distribution of individual level data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after closing baseline data collection with no end date
Access Criteria: Data will be shared in accordance with the NIH Helping to End Addiction Long-term (HEAL) Initiative Public Access and Data Sharing Policy. All data will be submitted to the NAHDAP repository and will be findable and accessible through the HEAL Initiative Data Ecosystem. All data will also be submitted to the NIDA-funded Methodology and Advanced Analytics Resource Center (MAARC) located at the University of Chicago, a data commons built for the purpose of sharing research data collected by research "hubs" within the NIDA-funded Justice Community Overdose Innovation Network (JCOIN). Data will be shared with investigators working under an institution with Federal Wide Assurance (FWA) and could be used for secondary study purposes. Requested primary study data and metadata (e.g., format and organization) will be made available to investigators according to the policies of the University of Chicago MAARC and the NAHDAP repository.
URL: https://grants.nih.gov/policy-and-compliance/policy-topics/sharing-policies/dms/policy-overview

REFERENCES:
- See also: Just Care for Families (JCFF) website — https://www.justcareforfamilies.org

DOCUMENTS (2):
  • Informed Consent Form: Guardian (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT07365293/ICF_000.pdf
  • Informed Consent Form: Participant (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT07365293/ICF_001.pdf